CLINICAL TRIAL: NCT04791059
Title: Low-dose S-ketamine and Dexmedetomidine in Combination With Opioids for Patient-controlled Analgesia After Scoliosis Correction Surgery: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Low-dose S-ketamine and Dexmedetomidine in Combination With Opioids for Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-465
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Scoliosis Correction; Postoperative Analgesia; S-ketamine; Dexmedetomidine; Sufentanil
Keywords: Scoliosis correction; Postoperative analgesia; S-ketamine; Dexmedetomidine; Sufentanil
MeSH Terms: interventions — Esketamine; Dexmedetomidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined analgesia group (Experimental): Patient-controlled analgesia is established with S-ketamine 50 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lock-out interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: S-ketamine; Drug: Dexmedetomidine; Drug: Sufentanil
- Control group (Placebo Comparator): Patient-controlled analgesia is established with sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lock-out interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: S-ketamine — S-ketamine 50 mg is included in the mixture for patient-controlled analgesia.
  Arms: Combined analgesia group
Drug: Dexmedetomidine — Dexmedetomidine 200 microgram is included in the mixture for patient-controlled analgesia.
  Arms: Combined analgesia group
Drug: Sufentanil — Sufentanil 4 microgram/kg (maximum 250 microgram) is included in the mixture for patient-controlled analgesia.

SUMMARY:
Scoliosis correction surgery is followed with severe pain. Patients after scoliosis correction surgery usually require high dose opioids and long duration analgesia, which may increase side effects and even drug tolerance. S-ketamine is the pure dextrorotatory enantiomer of ketamine with stronger analgesic effect and less side effects, but mental side effects is a major concern. Dexmedetomidine can be used as an analgesic supplement; it also improves sleep quality in postoperative patients. We hypothesize that low-dose ketamine and dexmedetomidine in combination with opioids may have synergistic effect in analgesia and reduce drug-related side effects. This study aims to explore the effect of low-dose of S-ketamine and dexmedetomidine in combination with opioids for postoperative patient-controlled intravenous analgesia in patients following scoliosis correction surgery.

DETAILED DESCRIPTION:
Scoliosis correction surgery is followed with severe pain. The reported median pain score on the first day after surgery is median 7 (IQR 4, 8); with an incidence of persistent postoperative pain from 5% to 75%. Most patients undergoing this surgery are young and adolescents; they are sensitive to pain and usually require higher dose analgesics and a long duration analgesia. The total dose of opioids required for postoperative analgesia is about 2-4 times higher than that after other surgeries. But even with high dose opioids, the analgesic effect remains unsatisfied. Furthermore, high dose opioids may cause side effects such as respiratory depression, drowsiness, nausea, vomiting, skin itching, and even drug tolerance.

Ketamine is a noncompetitive N-methyl-D-aspartate receptor antagonist (NMDA) with analgesic and anti-hyperalgesia effects. It is widely used for anesthesia induction in critically ill patients, pediatric anesthesia and postoperative analgesia. The advantages of ketamine include mild influence on respiratory and circulatory function, and good analgesic effect. Recent guidelines recommends the use of low-dose ketamine infusion for postoperative analgesia in patients with moderate to severe pain, in order to reduce the consumption of opioids. S-ketamine is the pure dextrorotatory enantiomer of ketamine with stronger analgesic effect and lower incidence of adverse reactions.

Dexmedetomidine is a highly selective α2 receptor agonist with effects of antianxiety, sedation and analgesia. When used as a supplement, it improves analgesic effect, and reduces opioid consumption and opioid related adverse reactions. In the same time, dexmedetomidine activates the endogenous sleep pathway and improves sleep quality by prolonging total sleep time, increasing sleep efficiency, and promoting subjective sleep quality.

It is worthy to note that ketamine can produce adverse reactions such as agitation, delirium and anxiety, and increase the incidence of hallucinations and nightmares when the given dose is slightly higher; whereas the sedative effect of dexmedetomidine may help to reduce the adverse effects of ketamine. We hypothesize that low-dose ketamine and dexmedetomidine in combination with opioids may have synergistic effects in postoperative analgesia and reduce drug-related adverse reactions.

This study aims to explore the effect of low-dose of S-ketamine and dexmedetomidine in combination with opioids for postoperative patient-controlled intravenous analgesia in patients following scoliosis correction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, body weight ≥ 40 kg;
* Scheduled to undergo scoliosis correction with pedicle screw fixation;
* Planned to use patient-controlled intravenous analgesia after surgery.

Exclusion Criteria:

* Refused to participate in the study;
* Preoperative sick sinus syndrome, severe sinus bradycardia (heart rate < 50 beats/min), atrioventricular block grade II or above without pacemaker; or comorbid with congenital heart disease, arrhythmia, or other serious cardiovascular diseases with a cardiac function grade ≥ III;
* Patients with obstructive sleep apnea syndrome, or a STOP-Bang score ≥ 3 in combination with a serum HCO3- level ≥ 28 mmol/L;
* History of hyperthyroidism and pheochromocytoma;
* History of schizophrenia, epilepsy, myasthenia gravis, or delirium;
* Severe liver dysfunction (child Pugh grade C), severe renal dysfunction (preoperative dialysis), or American Society of Anesthesiologists grade ≥ IV;
* Barrier in communication;
* Other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Percent of patients with moderate to severe pain within 72 hours | Up to 72 hours after surgery
  Pain severity is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) twice daily (8:00-10:00 and 18:00-20:00) at rest and with movement. Moderate to severe pain is defined as any NRS pain score of 4 or higher.

SECONDARY OUTCOMES:
NRS pain score (at rest and with movement) at various timepoints after surgery | Up to 72 hours after surgery
  Pain severity is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) twice daily (8:00-10:00 and 18:00-20:00) at rest and with movement. Moderate to severe pain is defined as any NRS pain score of 4 or higher.
Cumulative opioid consumption | Up to 72 hours after surgery
  Cumulative opioid consumption
Cumulative analgesic consumption | Up to 72 hours after surgery
  Cumulative analgesic consumption
Agitation and sedation score at various timepoints after surgery | Up to the 5th day after surgery
  Agitation and sedation score is evaluated with the Richmond Agitation and Sedation Scale (RASS, with scores ranging from -5 [unarousable] to +4 [combative] and 0 indicates alert and calm) twice daily (8:00-10:00 and 18:00-20:00).
Incidence of postoperative delirium within the first 5 days | Up to the 5th day after surgery
  Delirium is assessed with the Three-dimensional Confusion Assessment Method (3D CAM) twice daily (8:00-10:00 and 18:00-20:00).
Subjective sleep quality during the first 5 postoperative days | Up to the 5th day after surgery
  Subjective sleep quality is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = the best sleep and 10 = no sleep at all) once daily (8:00-10:00)
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Duration requiring analgesics within 30 days after surgery | Up to 30 days after surgery
  Duration requiring analgesics within 30 days after surgery
Incidence of postoperative complications within 30 days | Up to 30 days after surgery
  Postoperative complications are defined as new-onset medical conditions that were deemed harmful and required therapeutic intervention (i.e., grade II or higher on the Clavien-Dindo classification)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Hussain A, Erdek M. Interventional pain management for failed back surgery syndrome. Pain Pract. 2014 Jan;14(1):64-78. doi: 10.1111/papr.12035. Epub 2013 Feb 3. PMID 23374545
- [Background] Seki H, Ideno S, Ishihara T, Watanabe K, Matsumoto M, Morisaki H. Postoperative pain management in patients undergoing posterior spinal fusion for adolescent idiopathic scoliosis: a narrative review. Scoliosis Spinal Disord. 2018 Sep 12;13:17. doi: 10.1186/s13013-018-0165-z. eCollection 2018. PMID 30214945
- [Background] Nielsen RV. Adjuvant analgesics for spine surgery. Dan Med J. 2018 Mar;65(3):B5468. PMID 29510816
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Focus (Am Psychiatr Publ). 2019 Jan;17(1):55-65. doi: 10.1176/appi.focus.17105. Epub 2019 Jan 7. PMID 32015715
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Stone LS, MacMillan LB, Kitto KF, Limbird LE, Wilcox GL. The alpha2a adrenergic receptor subtype mediates spinal analgesia evoked by alpha2 agonists and is necessary for spinal adrenergic-opioid synergy. J Neurosci. 1997 Sep 15;17(18):7157-65. doi: 10.1523/JNEUROSCI.17-18-07157.1997. PMID 9278550
- [Background] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Gao Y, Deng X, Yuan H, Leng Y, Zhang T, Xu X, Tian S, Fang J, Ouyang W, Wu X. Patient-controlled Intravenous Analgesia With Combination of Dexmedetomidine and Sufentanil on Patients After Abdominal Operation: A Prospective, Randomized, Controlled, Blinded, Multicenter Clinical Study. Clin J Pain. 2018 Feb;34(2):155-161. doi: 10.1097/AJP.0000000000000527. PMID 28654556
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Meng ZT, Cui F, Li XY, Wang DX. Epidural morphine improves postoperative analgesia in patients after total knee arthroplasty: A randomized controlled trial. PLoS One. 2019 Jul 1;14(7):e0219116. doi: 10.1371/journal.pone.0219116. eCollection 2019. PMID 31260468
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Derived] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963